CLINICAL TRIAL: NCT03372681
Title: A Superiority Study for Postoperative Reflux After Distal Gastrectomy With Antiperistaltic vs Isoperistaltic Billroth II + Braun Anastomosis
Brief Title: Comparative Study of Antiperistaltic vs Isoperistaltic Billroth II + Braun Anastomosis for Postoperative Reflux
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShanghaiMISC-B2+Braun
Record Dates: First submitted 2017-12-10; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Gastric Cancer; Postoperative Complications
Keywords: Distal Gastrectomy; Postoperative Reflux Rate; Gastric Cance; Laparoscopic Surgery
MeSH Terms: conditions — Stomach Neoplasms; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antiperistaltic (Experimental): In this group patients undergo the distal gestrectomy with antiperistaltic Billroth II + Braun anastomosis
  Interventions: Procedure: Antiperistaltic Billroth II + Braun anastomosis
- Isoperistaltic (Active Comparator): In this group patients undergo the distal gestrectomy with isoperistaltic Billroth II + Braun anastomosis
  Interventions: Procedure: Isoperistaltic Billroth II + Braun anastomosis

INTERVENTIONS:
Procedure: Isoperistaltic Billroth II + Braun anastomosis — Laparoscopic distal gestrectomy will be applied with Isoperistaltic Billroth II + Braun reconstruction
  Arms: Isoperistaltic
Procedure: Antiperistaltic Billroth II + Braun anastomosis — Laparoscopic distal gestrectomy will be applied with antiperistaltic Billroth II + Braun reconstruction
  Arms: Antiperistaltic

SUMMARY:
Postoperative gastroesophageal reflux is one of the most common complications of distal gastrectomy. With more attention paid on it by surgeons, several new operation methods have been practised. Among all these, distal gastrctomy with Billroth II + Braun anastomosis was reported to be an useful method to decrease postoperative reflux rate. Meanwhile, the direction of anastomotic peristalsis has also been reported to affect the anastomosis and thus make difference in reflux rate. We design this study to investigate the potential effect and the superiority of antiperistaltic vs isoperistaltic Billroth II + Braun reconstruction in distal gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed as gastric cancer before surgery
* Clinical staging: cT1-4aN0-3M0
* Postoperative evaluation concluded B-II B anastomosis
* Consent assigned

Exclusion Criteria:

* Diagnosed with other malignancies within 2 years
* Gastric cancer with clinical staging: cT4b or M1
* Women with pregnancy or breast-feeding
* Emergency procedures
* Consent not assigned

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Reflux Rate | 1 yrs
  The rate of bile reflux within 1yrs postoperation

SECONDARY OUTCOMES:
Disease-free survival | 3yrs
  3yrs DFS
Overall survival | 3 yrs
  3yrs OS
Surgery-related reflux gastritis rate | 1yrs
  The rate of surgery-related reflux gastritis rate
Surgery-related reflux esophagitis rate | 1 yrs
  The rate of surgery-related reflux esophagitis rate

CONTACTS AND LOCATIONS:
Overall Officials: Minhua Zheng, M.D. PhD., Study Director — MISC, Ruijin Hospital, School of Medicine, Shanghai Jiao Tong University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cui LH, Son SY, Shin HJ, Byun C, Hur H, Han SU, Cho YK. Billroth II with Braun Enteroenterostomy Is a Good Alternative Reconstruction to Roux-en-Y Gastrojejunostomy in Laparoscopic Distal Gastrectomy. Gastroenterol Res Pract. 2017;2017:1803851. doi: 10.1155/2017/1803851. Epub 2017 Jan 9. PMID 28163716
- [Background] In Choi C, Baek DH, Lee SH, Hwang SH, Kim DH, Kim KH, Jeon TY, Kim DH. Comparison Between Billroth-II with Braun and Roux-en-Y Reconstruction After Laparoscopic Distal Gastrectomy. J Gastrointest Surg. 2016 Jun;20(6):1083-90. doi: 10.1007/s11605-016-3138-7. Epub 2016 Apr 11. PMID 27067234